CLINICAL TRIAL: NCT06736210
Title: The Role of Muscle Elastic Properties of Extrinsic Foot Muscles, Muscle Oxygenation and Plantar Pressure Change in Determining Diabetic Foot Ulcer Risk
Brief Title: The Role of Extrinsic Foot Muscles Chances in Determining the Risk of Diabetic Foot Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Ali Ilez, Research Assistant, Istanbul Saglik Bilimleri University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: SBU-FTR-AI-01
Record Dates: First submitted 2024-12-10; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Foot; Diabetes Mellitus
Keywords: Diabetic Foot; Muscle Oxygenation; Muscle Elasticity
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Health Control Group (Experimental): The healthy control group consisted of 10 participants with no history of foot or ankle injuries or systemic diseases, ensuring a baseline for comparison. Assessments included isokinetic testing for plantar flexor (PF) and dorsiflexor (DF) muscle strength and endurance at angular velocities of 30°/s and 120°/s, respectively. Additionally, functional evaluations such as the physical performance (heel-rise) test and patient-reported outcome measures (AOFAS and FAOS scores) were conducted. These evaluations provided a comprehensive understanding of muscle performance and functional status in healthy individuals, serving as a reference point for interpreting deviations observed in the Lisfranc injury group.
  Interventions: Other: Muscle Elastic Properties Measurement; Other: Muscle Oxygen Saturation (SmO2); Other: Plantar Pressure Analysis
- IWDGF-0 (Experimental): The IWGDF 0 group included 10 patients classified as having no immediate risk for diabetic foot ulcers. Assessments focused on evaluating the biomechanical and functional parameters of extrinsic foot muscles. Muscle elasticity and dynamic stiffness were measured using the MyotonPro device, while muscle oxygenation levels (SmO2) were recorded pre- and post-exercise using the MOXY device. Plantar pressure analysis was performed under both static and dynamic conditions to identify subtle variations in pressure distribution and foot biomechanics. These evaluations aimed to detect early indicators of potential foot complications, even in patients without apparent risk, providing critical data for preventive strategies.
  Interventions: Other: Muscle Elastic Properties Measurement; Other: Muscle Oxygen Saturation (SmO2); Other: Plantar Pressure Analysis
- IWDGF-1 (Experimental): The IWGDF 1 group comprised 10 patients identified as having low risk for diabetic foot ulcers. Comprehensive assessments were conducted to evaluate the biomechanical and functional properties of their extrinsic foot muscles. Elasticity and dynamic stiffness of the tibialis anterior, gastrocnemius medialis, gastrocnemius lateralis, and peroneus longus muscles were measured using the MyotonPro device. Muscle oxygenation levels (SmO2) were monitored pre- and post-exercise using the MOXY device to determine oxygen utilization and recovery capacity. Additionally, plantar pressure was analyzed under static and dynamic conditions to assess changes in pressure distribution and foot biomechanics. These detailed evaluations highlighted early biomechanical and functional changes, emphasizing the importance of targeted interventions in this low-risk group to prevent progression to higher risk categories.
  Interventions: Other: Muscle Elastic Properties Measurement; Other: Muscle Oxygen Saturation (SmO2); Other: Plantar Pressure Analysis

INTERVENTIONS:
Other: Muscle Elastic Properties Measurement — Using the MyotonPro device, the elastic properties, including stiffness, elasticity, and tone, were evaluated for the tibialis anterior, gastrocnemius medialis, gastrocnemius lateralis, and peroneus longus muscles. Measurements were performed in a controlled laboratory setting.
Other: Muscle Oxygen Saturation (SmO2) — Muscle oxygenation levels were measured before and after a standardized exercise protocol using the MOXY device. The exercise protocol consisted of a light-intensity dynamic task tailored to minimize fatigue and mimic functional activity.
Other: Plantar Pressure Analysis — Plantar pressure was assessed both statically and dynamically using a pressure-mapping platform. This provided data on pressure distribution, contact times, and high-pressure areas across the foot during various conditions.

SUMMARY:
Many foot and lower limb disorders resulting from diabetes, such as deformity, muscle weakness, reduced range of motion, stiffness of connective tissue, amount of oxygenation, functional capacity, poor balance and coordination, can potentially be corrected or prevented with specific interventions (15). It is important to diversify assessment methods for the development and elaboration of prevention strategies. Rapid, low-cost and detailed evaluations provide good planning of treatment. According to the International Diabetic Foot Study Group (IDFG) scale used to determine the risk of diabetic foot ulcer, it is thought that performing a plantar pressure analysis of a patient with diabetes to determine the people who do not have foot ulcers but are at risk, knowing the difference in the amount of muscle oxygenation of the muscles around the foot and ankle with healthy people and the change in muscle elastic properties will be important in terms of preventing the occurrence of diabetic foot ulcers and determining the changes of the treatments applied in the lower extremities.

DETAILED DESCRIPTION:
Recent guidelines for the treatment and prevention of diabetic foot complications emphasize the management/control of diabetes, foot care, patient education and self-management of foot care . Other rehabilitation approaches, including exercise therapy, have recently come to the forefront in the literature within the scope of preventive treatments. Exercises have been shown to be beneficial in diabetic patients, especially in increasing nerve velocity conduction in the lower extremities . As a result of these recommendations, evaluation of the risk of diabetic foot ulceration before ulceration develops, detailed analysis of all tissues and systems expected to be affected may be solved with preventive strategies by reducing the need for treatment.

The change in plantar pressure distribution in patients with diabetes is one of the mechanisms that form the basis of the mechanisms of foot ulcer formation. Altered biomechanical structure, high intensity and repetitive diffuse pressure due to neuropathy, and insufficiency of vascular tissues caused by peripheral arterial disease directly affect the plantar pressure distribution . Determining this change before diabetic wound formation, analyzing the changing plantar pressure ratios and determining the condition in the presence of neuropathy may improve the quality of the treatment program to be created.

In the study conducted by Stephens et al. In the study conducted by Stephens et al. the plantar surface tissue of the intrinsic foot muscles oxidized following exercise interventions in patients diagnosed with diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria for Patients with Diabetes:

* Willingness to participate in the study
* Absence of current or past diabetic foot ulcers
* Classification within the 0 or 1 categories of the IWGDF classification system

Inclusion Criteria for Sedentary Healthy Participants:

* Willingness to participate in the study
* Not engaging in active sports activities
* Absence of current or past foot ulcers

Exclusion Criteria for all group:

* Presence of orthopedic, musculoskeletal, vestibular, visual, or neurological problems affecting mobility (other than DPN)
* History of prior orthopedic surgical intervention in the lower extremity
* Dementia or inability to provide consistent information
* Presence of major vascular complications (venous or arterial ulcers)
* Diagnosis of PAH (Peripheral Arterial Hypertension)
* Presence of plantar ulcers during or prior to the assessment
* Inability to walk independently without pain or assistive devices
* Illiteracy
* Presence of any foot deformity

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Muscle Elastic Properties | Measured within a 1-month period.
  Stiffness, elasticity, and tone of the tibialis anterior, gastrocnemius medialis, gastrocnemius lateralis, and peroneus longus muscles measured using the MyotonPro device.
  Key Metrics: Differences in muscle stiffness, tone, and elasticity between groups.

SECONDARY OUTCOMES:
Muscle Oxygenation (SmO2) | Measured within a 1-month period.
  Changes in local oxygen saturation (SmO2) levels of the targeted muscles, measured pre- and post-exercise using the MOXY device.
  Comparison of SmO2 levels between IWGDF 0, IWGDF 1, and healthy control groups. Key Metrics: Reduction in SmO2 levels and recovery trends post-exercise
Plantar Pressure Parameters | Measured within a 1-month period.
  Static and dynamic plantar pressure analysis to identify high-pressure regions and foot loading patterns.
  Key Metrics:
  Average plantar pressure values in midfoot and forefoot regions. Contact times and pressure distribution in dynamic gait analysis.

OTHER OUTCOMES:
Functional Integration | Measured within a 1-month period.
  Evaluation of the relationship between plantar pressure patterns and muscle biomechanical properties across all groups.

CONTACTS AND LOCATIONS:
Overall Officials: Defne KAYA UTLU, PhD, Study Director — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences Physical Therapy and Rehabilitation Lab, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Armstrong DG, Tan TW, Boulton AJM, Bus SA. Diabetic Foot Ulcers: A Review. JAMA. 2023 Jul 3;330(1):62-75. doi: 10.1001/jama.2023.10578. PMID 37395769